CLINICAL TRIAL: NCT05490173
Title: The Pilot Experimental Study of the Neuroprotective Effects of Exosomes in Extremely Low Birth Weight Infants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal State Budget Institution Research Center for Obstetrics, Gynecology and Perinatology Ministry of Healthcare (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ncagp4382277
Record Dates: First submitted 2022-07-04; First posted 2022-08-05 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Premature Birth; Extreme Prematurity; Preterm Intraventricular Hemorrhage; Hypoxia-Ischemia, Cerebral; Neurodevelopmental Disorders
Keywords: Extremely low birth weight, neuroprotection
MeSH Terms: conditions — Premature Birth; Hypoxia-Ischemia, Brain; Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: Participants (ELBW infants GA 25/0-27/6 week) are randomized to one of two groups in parallel for the duration of the study. The first group (exosome treatment group) will receive intranasal administration of exosomes and the second (control group) will not receive exosomes. Patients in both groups will receive standard basic therapy
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal exosomes administration (Experimental): ELWB newborns who will receive intranasal exosomes
  Interventions: Other: Exosomes derived from mesenchymal stromal cells (MSCs)
- Control (No Intervention): ELWB newborns who will not receive intranasal exosomes

INTERVENTIONS:
Other: Exosomes derived from mesenchymal stromal cells (MSCs) — Exosomes derived from mesenchymal stromal cells (MSCs) will be administered intranasal in ELBW infants
  Arms: Intranasal exosomes administration

SUMMARY:
To study the safety and efficacy of intranasal administration of exosomes derived from mesenchymal stromal cells on long-term neurodevelopmental outcome in extremely low birth weight infants born at gestational age 25/0-27/6 weeks.

DETAILED DESCRIPTION:
Surviving extremely low birth weight (ELBW) infants are at risk of severe neurodevelopmental disability. Exosomes or extracellular vesicles (EVs) derived from mesenchymal stromal cells (MSCs) can mediate a variety of different effects, including synaptic plasticity, nutritional metabolic support, nerve regeneration, inflammatory response, anti-stress effect, cellular waste disposal, treating neurological injury, preventing hemorrhagic and ischemic brain lesions, playing an important role in health and neuroprotection in extremely premature newborns during neonatal intensive care.

The proposed blinded randomized controlled trial was designed to compare the effect of intranasal administration of exosomes on long-term neurodevelopmental outcome in ELBW infants.

ELBW infants will be randomized to receive (group 1) and not receive exosomes (control group).

Group 1 - Neonates will receive exosomes (1 dose will be obtained from a daily conditioned culture medium of 120 million MSCs) suspended in 500 µl of phosphate buffer in each nostril at 50 µl with an interval of 2-3 minutes. The therapeutic course will consist of 5 instillations with an interval of 1 days.

The primary outcome measure is the incidence of death, the incidence of survival with any of either severe intraventricular hemorrhage (IVH), cystic periventricular leukomalacia (PVL), or brain injury on cranial ultrasound and MRI or major neurodevelopmental impairment determined at 36 months of age corrected for prematurity (where major neurodevelopmental impairment is defined as any of the following: cognitive deficit, cerebral palsy, or severe visual or hearing impairment. Cognitive delay defined as mental developmental index (MDI) score of the Griffiths-II and Bayley Scales of Infant Development (2nd edition) < 85, cerebral palsy, or severe visual or hearing impairment.

To investigate this outcomes and the mechanisms by which extracellular vesicles (EVs) might effect we will analyze the biomarkers of perinatal brain injury (S-100, NSE, EPO) and mRNA.

Key secondary outcomes are incidences of short term outcomes: individual components of the composite primary outcome, survival with and without major neonatal morbidity including severe retinopathy of prematurity (ROP), bronchopulmonary dysplasia (BPD), necrotizing enterocolitis (NEC).

Safety analyses will assess the injures or damages of the nasal mucosa, allergic reaction to EVs and any adverse events after intranasal administration of EVs.

The results of this trial may help to improve the quality of life of ELBW infants and reduce long-term health care costs.

ELIGIBILITY:
Inclusion Criteria:

• Premature newborns of gestational age (GA) 25/0-27/6 weeks,

Exclusion Criteria:

* Missing written parental consent
* Damages to the nasal mucosa
* Maxillofacial defects
* Major congenital anomalies (including chromosomal aberrations, cyanotic congenital heart defects, syndromes likely affecting long-term outcome, and major congenital malformations requiring surgical correction during newborn period)
* Infants who died before 48 hours, infants in whom the clinical decision to withhold intensive care was made, infants who were not considered viable
* Infants with edematous hemolytic disease of newborns, non-immune fetal dropsy,
* Multifetal Gestations
* Participation in another study with ongoing use of an unlicensed investigational product from 28 days before study enrollment until the end of the study

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2022-10-05 (Estimated); Primary Completion 2026-05-22 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Occurrence and rate of dose limiting toxicity | Up to 1 week following after intranasal administration of EVs
  Dose limiting toxicity consists of the following events:
  Death occurring within 24 hours after intranasal administration of EVs; Hypersensitivity / anaphylactic to EVs defined as any severe systemic inflammatory response syndrome with negative blood culture not consistent with the overall clinical course of the infant occurring within 72 hours after intranasal administration of EVs; Any other serious adverse event not expected in this patient population for which there is no alternative explanation but the administration of EVs, occurring within 1 week of injection.

SECONDARY OUTCOMES:
Rate of death | From enrollment until discharge or 40 weeks corrected gestational age (whichever occurs first)
  Rate of death until discharge or 40 weeks corrected gestational age, whichever comes first
Occurrence of Other Severe Complications of Prematurity | From enrollment until discharge or 40 weeks corrected gestational age (whichever occurs first)
  * Blood culture-proven sepsis
  * Patent ductus arteriosus (treated medically or surgically)
  * Necrotizing enterocolitis
  * Isolated intestinal perforation
  * Retinopathy of prematurity requiring treatment
  * Severe intraventricular hemorrhage (≥ grade 3)
  * Cystic periventricular leukomalacia
  * Incidence and Severity of BPD, Measured as mild, moderate, or severe
Need for Ventilatory Support | From enrollment until discharge, 40 weeks corrected gestational age, or death (whichever occurs first)
  * Time to extubation
  * Duration of mechanical ventilation
  * Duration of non-invasive positive pressure respiratory support
  * Duration of supplemental oxygen
Changes in Hemodynamics | Time Frame: At enrollment, 48 hours following intranasal administration of EVs, 28 days of life, and 36 weeks corrected gestational age
  Targeted neonatal echocardiography to assess
Feasibility: Administration | Day of life 1-10
  Successful recruitment and administration of extracellular vesicles to 10 patients in 18 months
Feasibility: Recruitment Efficiency | Day of life 1-10
  * Proportion of potentially eligible patients that are successfully screened
  * Proportion of participants successfully screened who do not enroll (reason for failure to enroll will be recorded)
Feasibility: Recruitment Timing | Day of life 1-10
  * Median time from screening to enrollment
  * Median time from screening to extracellular vesicles
Feasibility: Participant Retainment | From enrollment until follow-up at 18-36 months-of-age
  * Proportion of patients that do not complete administration of extracellular vesicles
  * Proportion of patients enrolled that do not undergo scheduled follow-up
Griffiths-II and Bayley Scales of Infant Development (2nd edition) | 18-36 months-of-age
  Assessment of cognitive, language, and motor development. Cognitive delay defined as mental developmental index (MDI) score of the Griffiths-II and Bayley Scales of Infant Development (2nd edition) < 85, cerebral palsy, or severe visual or hearing impairment.
Long-term Safety Follow-Up | 3 years following follow-up visit
  Participant's overall health will be assessed through a questionnaire administered over the phone, once a year for 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Ionov, PhD, MD, Principal Investigator — NATIONAL MEDICAL RESEARCH CENTER FOR OBSTETRICS, GYNECOLOGYAND PERINATOLOGY NAMED AFTER ACADEMICIAN V.I.KULAKOV; Ekaterina Balashova, PhD, MD, Principal Investigator — NATIONAL MEDICAL RESEARCH CENTER FOR OBSTETRICS, GYNECOLOGYAND PERINATOLOGY NAMED AFTER ACADEMICIAN V.I.KULAKOV; Denis Silachev, PhD, MD, Principal Investigator — NATIONAL MEDICAL RESEARCH CENTER FOR OBSTETRICS, GYNECOLOGYAND PERINATOLOGY NAMED AFTER ACADEMICIAN V.I.KULAKOV; Anna Kirtbaya, PhD, MD, Principal Investigator — NATIONAL MEDICAL RESEARCH CENTER FOR OBSTETRICS, GYNECOLOGYAND PERINATOLOGY NAMED AFTER ACADEMICIAN V.I.KULAKOV; Victor Zubkov, PhD, MD, Principal Investigator — NATIONAL MEDICAL RESEARCH CENTER FOR OBSTETRICS, GYNECOLOGYAND PERINATOLOGY NAMED AFTER ACADEMICIAN V.I.KULAKOV; Dmitriy Degtyarev, PhD, MD, Principal Investigator — NATIONAL MEDICAL RESEARCH CENTER FOR OBSTETRICS, GYNECOLOGYAND PERINATOLOGY NAMED AFTER ACADEMICIAN V.I.KULAKOV
Locations (1):
- Federal State Budget Institution Research Center for Obstetrics, Gynecology and Perinatology Ministry of Healthcare, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ophelders DR, Wolfs TG, Jellema RK, Zwanenburg A, Andriessen P, Delhaas T, Ludwig AK, Radtke S, Peters V, Janssen L, Giebel B, Kramer BW. Mesenchymal Stromal Cell-Derived Extracellular Vesicles Protect the Fetal Brain After Hypoxia-Ischemia. Stem Cells Transl Med. 2016 Jun;5(6):754-63. doi: 10.5966/sctm.2015-0197. Epub 2016 May 9. PMID 27160705
- [Background] Drommelschmidt K, Serdar M, Bendix I, Herz J, Bertling F, Prager S, Keller M, Ludwig AK, Duhan V, Radtke S, de Miroschedji K, Horn PA, van de Looij Y, Giebel B, Felderhoff-Muser U. Mesenchymal stem cell-derived extracellular vesicles ameliorate inflammation-induced preterm brain injury. Brain Behav Immun. 2017 Feb;60:220-232. doi: 10.1016/j.bbi.2016.11.011. Epub 2016 Nov 12. PMID 27847282
- [Result] Gamage TKJB, Fraser M. The Role of Extracellular Vesicles in the Developing Brain: Current Perspective and Promising Source of Biomarkers and Therapy for Perinatal Brain Injury. Front Neurosci. 2021 Sep 24;15:744840. doi: 10.3389/fnins.2021.744840. eCollection 2021. PMID 34630028
- See also: The Role of Extracellular Vesicles in the Developing Brain: Current Perspective and Promising Source of Biomarkers and Therapy for Perinatal Brain Injury — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC8498217/
- See also: The Role of Extracellular Vesicles in the Developing Brain: Current Perspective and Promising Source of Biomarkers and Therapy for Perinatal Brain Injury — http://pubmed.ncbi.nlm.nih.gov/34630028/
- See also: Mesenchymal Stromal Cell-Derived Extracellular Vesicles Protect the Fetal Brain After Hypoxia-Ischemia — http://pubmed.ncbi.nlm.nih.gov/27160705/
- See also: Mesenchymal stem cell-derived extracellular vesicles ameliorate inflammation-induced preterm brain injury — http://pubmed.ncbi.nlm.nih.gov/27847282/